CLINICAL TRIAL: NCT05884424
Title: Effectiveness and Cost-Effectiveness of Robot Therapy With the Paro Robot in People Living With Dementia: A Randomized Controlled Multicenter Clinical Trial
Brief Title: Effectiveness and Cost-Effectiveness of Robot Therapy With the Paro Robot in People Living With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Mayores y Servicios Sociales (IMSERSO) (Other Government)
Collaborators: Asturhealth SL (Unknown); Servicio de Evaluación y Planificación del Servicio Canario de la Salud (SESCS) (Unknown)
Responsible Party: Principal Investigator, Enrique Perez Saez, Neuropsychologist, Instituto de Mayores y Servicios Sociales (IMSERSO)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/22
Record Dates: First submitted 2023-04-14; First posted 2023-06-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Dementia; Neurocognitive Disorders; Mild Cognitive Impairment
Keywords: Dementia; Neurocognitive Disorders; Mild Cognitive Impairment; Robot therapy; Quality of life; Neuropsychiatric symptoms; Older adult; Robot; Cost-effectiveness
MeSH Terms: conditions — Dementia; Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The investigators propose the conduct of a randomized and controlled multicenter pragmatic clinical trial to compare 12 weeks of robot therapy sessions with the PARO robot versus 12 weeks of standard care. Participants who meet the inclusion criteria will be allocated by block randomization to either the PARO robot intervention group or the standard care control group. Participants allocated to the PARO group will undergo three intervention sessions per week for 12 weeks, in addition to continuing their standard care. Participants in the control group will maintain their standard care, participating in those activities previously assigned in their individual care plan. In addition, follow-up will be performed 12 weeks after the end of the intervention to assess the duration of the effects.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The technician in charge of assessing users participating in the study must be blinded throughout the intervention, i.e., he/she will not be able to know whether the assessed users belong to the experimental group or to the control group.
  The person from CREA - Imserso in charge of randomization and data analysis will also be blinded.
  The participants and the technician implementing the intervention cannot be blinded, due to the inherent nature of the intervention.
  Data analysis will also be performed blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARO Therapy Robot (Experimental): Participants allocated to the PARO Therapy Robot group will undergo three group robot therapy sessions per week for 12 weeks, in addition to continuing their standard care.
  Interventions: Behavioral: PARO Therapy Robot
- Control (No Intervention): Participants in the control group will maintain their standard care, participating in those activities previously assigned in their individual care plan.

INTERVENTIONS:
Behavioral: PARO Therapy Robot — Participants allocated to the PARO Therapy Robot group will receive three group robot therapy sessions per week for 12 weeks, in addition to continuing their standard care.
  Robot therapy session will last 20 minutes. The sessions will be partially guided, intending to allow participants to interact with the robot seal freely for as long as possible, but redirecting the activity if necessary. The sessions will be conducted in group format, in groups of 4 users, with participants sitting in a circle around a table. The professional conducting the sessions will be a therapist with experience in NPT for people living with dementia, and who has attended the training session on the study intervention protocol.
  The sessions will be structured as follows:
  1. Welcome and presentation.
  2. Main activity with PARO.
  3. PARO cleaning.
  4. End of session. A total of 13 different sessions are proposed, to be conducted in a cyclical manner (each session 3 times, except sessions 1 and 2).
  Other Names: PARO
  Arms: PARO Therapy Robot

SUMMARY:
The purpose of this study is to evaluate the effectiveness and cost-effectiveness of group robot therapy with the PARO therapy robot in terms of quality of life and neuropsychiatric symptoms in people living with dementia in residential centers. In addition, the acceptability of the robot on the part of the users participating in the study will be evaluated.

The evaluation will be carried out through a multicenter pragmatic clinical trial randomized to an intervention group (PARO therapy robot) or a control group (treatment as usual). Participants in the intervention group will complete three sessions per week with the PARO therapy robot during 12 weeks. Participants in the control group will maintain their standard care. In addition, a follow-up evaluation will be made three months after the end of the intervention to assess the duration of the possible effects.

DETAILED DESCRIPTION:
The increase in life expectancy in recent decades has been associated with inevitable aging of the population and a rise in the prevalence of dementia. The World Health Organization (WHO) defines dementia as an acquired condition involving multiple cognitive disabilities that are sufficient to interfere with the daily life of the patients and their environment, with important associated personal suffering and economic costs. Despite advances in recent years, the diagnosis and course of dementia remains a challenge for professionals, and there continue to be important social and healthcare shortcomings regarding prevention, treatment and care.

Due to the deficiencies of the existing drugs, non-pharmacological therapies (NPT) are particularly relevant in the management of dementia. A NPT is any non-chemical, theoretically supported, focused and replicable intervention that is potentially able to produce a relevant benefit. Among these NPT, mention must be made of robot therapy, which involves the use of robots that simulate animals and are equipped with artificial intelligence and multiple sensors that allow them to behave and interact with users as if they were a real animal.

Therapy robots are regarded as an alternative to animal-assisted therapy, avoiding complications arising from the presence of animals while affording similar effects. The Personal Assistant Robot (PARO) robot seal was developed with this purpose in mind. It is the most widely used robot in the field of dementia, and also the most widely studied robot. Designed in Japan by Professor T. Shibata, PARO is an interactive robot with five types of sensors (light, touch, posture, temperature and sound), and it has demonstrated the ability to provide social and emotional stimulation.

In people living with dementia, robot therapy has been shown to offer psychological benefits (improved relaxation and motivation), physiological benefits (improved vital signs) and social benefits (stimulation of communication). In addition, the most recent studies have shown robot therapy to exert positive effects upon cognitive function, agitation, anxiety, depression, other neuropsychiatric symptoms and quality of life. However, other reviews have not recorded sufficient evidence of the positive effects of robot therapy upon cognition, neuropsychiatric symptoms or quality of life. Further quality studies are therefore needed on the effect of robot therapy in people living with dementia.

In this regard, the proposed study is aimed at evaluating the effectiveness and cost-effectiveness of group robot therapy intervention with the PARO robot in terms of quality of life and neuropsychiatric symptoms in people living with dementia in residential centers. In addition, the acceptability of the intervention on the part of the users participating in the study will be evaluated. For this purpose, a multicenter study will be carried out in the form of a randomized clinical trial in which the selected participants will be randomized to an intervention group (PARO Therapy Robot) or a control group (standard care).

Hypothesis:

* After the intervention, participants in the experimental group will improve their quality of life scores compared with the control group receiving standard care, where scores will be maintained or will get worse.
* Participants in the experimental group will have fewer neuropsychiatric alterations than participants in the control group.
* Participants in the experimental group will reduce their depression scores versus participants in the control group.
* Participants in the experimental group will experience less agitation than participants in the control group.
* Participants in the experimental group will experience less apathy than participants in the control group.
* The PARO robot will be well accepted by the individuals living with dementia.
* PARO Therapy Robot will be efficient in comparison with standard care. Objectives

The primary study objective is:

• To compare the effectiveness of the PARO Therapy Robot and standard care in improving the quality of life of people with dementia living in residential centers.

The secondary objectives are:

* To compare the effectiveness of the PARO Therapy Robot and standard care in reducing neuropsychiatric disorders in people with dementia. Specifically, efficacy will be compared in terms of:

  * Reducing depressive symptoms.
  * Reducing agitation.
  * Reducing apathy.
* To evaluate the acceptability of the PARO robot on the part of the patients.
* To perform a cost-effectiveness and cost-utility analysis, comparing the direct costs of the PARO Therapy Robot and standard care with the results afforded by the two alternatives.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the sites participating in the study.
* Persons over 60 years of age.
* A diagnosis of mild to moderate dementia (of any type) (Mini-Mental State Examination [MMSE] score between 13-25).
* Patients who have not previously participated in intervention sessions with the PARO robot and who do not participate in other robotic or animal-assisted interventions during the course of the study.
* Signing of informed consent by the person with dementia or the legal guardian.
* No firm and obvious rejection of the PARO therapy robot.

Exclusion Criteria:

* Presence of sensory limitations that preclude participation in the sessions.
* Health issues that advise against or impede participation in the sessions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | Baseline (T0)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | 12 weeks after the beginning of the intervention (T1)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.
Change in quality of life evaluated through Quality of Life - Alzheimer's Disease (QoL-AD) | 12 weeks after end of the intervention (T2)
  Quality of Life - Alzheimer's Disease (QoL-AD). QoL-AD is used to assess quality of life in people with dementia, based on the information provided by the patient (patient version). It consists of 13 items referring to perceived health status, mood, functional capacity, personal and leisure relationships, capacity to decide, and personal life as a whole. Each item is answered on a Likert-type scale from 1 (poor) to 4 (excellent). The score range from 13-52. Higher scores indicate better quality of life. This tool has good psychometric properties, and its use has been recommended by a European consensus to assess psychosocial interventions. The Spanish adaptation of this scale will be used.
Quality of life evaluated through EQ-5D-5L | Baseline (T0)
  EQ-5D-5L. The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way we have an index that can be used directly or combined with life years to calculate QALYs (quality-adjusted life years).
Change in quality of life evaluated through EQ-5D-5L | 12 weeks after the beginning of the intervention (T1)
  EQ-5D-5L. The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way we have an index that can be used directly or combined with life years to calculate QALYs (quality-adjusted life years).
Change in quality of life evaluated through EQ-5D-5L | 12 weeks after end of the intervention (T2)
  EQ-5D-5L. The EQ-5D-5L is a generic instrument for the assessment of health-related quality of life that can be used in both relatively healthy individuals and in groups of patients with different disease conditions. The individual evaluates his or her own state of health first as severity levels by dimensions (mobility, self-care, daily activities, pain/discomfort and anxiety/depression), and then using a more general evaluation visual analog scale (VAS). A third element is the social values index that is obtained for each health status generated by the instrument. The index ranges from 1 (best health status) to 0 (death), though there are negative values for the index, corresponding to those health statuses that are assessed as being worse than death. In this way we have an index that can be used directly or combined with life years to calculate QALYs (quality-adjusted life years).

SECONDARY OUTCOMES:
Mood assessed through the Geriatric Depression Scale-15 (GDS-15) | Baseline (T0)
  Geriatric Depression Scale (GDS-15). GDS-15 consists of 15 yes/no questions and the score ranges from 0-15. Scores of 6 or higher on a maximum of 15 points are considered to be indicative of depression. The Spanish adaptation of this scale will be used. This scale is administered to the person with dementia.
Change in mood assessed through the Geriatric Depression Scale-15 (GDS-15) | 12 weeks after the beginning of the intervention (T1)
  Geriatric Depression Scale (GDS-15). GDS-15 consists of 15 yes/no questions and the score ranges from 0-15. Scores of 6 or higher on a maximum of 15 points are considered to be indicative of depression. The Spanish adaptation of this scale will be used. This scale is administered to the person with dementia.
Change in mood assessed through the Geriatric Depression Scale-15 (GDS-15) | 12 weeks after end of the intervention (T2)
  Geriatric Depression Scale (GDS-15). GDS-15 consists of 15 yes/no questions and the score ranges from 0-15. Scores of 6 or higher on a maximum of 15 points are considered to be indicative of depression. The Spanish adaptation of this scale will be used. This scale is administered to the person with dementia.
Apathy assessed through the Apathy in Dementia-Nursing Home (APADEM-NH) | Baseline (T0)
  APADEM-NH explores the dimensions of thought deficit (33 items), emotional blunting (17 items), and cognitive inertia (16 items), based on a Likert-type scale from 0 (no apathy) to 3 (severe apathy). This scale will be completed by a regular caregiver of the person with dementia, who in this case will be a professional at the site.
Change in apathy assessed through the Apathy in Dementia-Nursing Home (APADEM-NH) | 12 weeks after the beginning of the intervention (T1)
  APADEM-NH explores the dimensions of thought deficit (33 items), emotional blunting (17 items), and cognitive inertia (16 items), based on a Likert-type scale from 0 (no apathy) to 3 (severe apathy). This scale will be completed by a regular caregiver of the person with dementia, who in this case will be a professional at the site.
Change in apathy assessed through the Apathy in Dementia-Nursing Home (APADEM-NH) | 12 weeks after end of the intervention (T2)
  APADEM-NH explores the dimensions of thought deficit (33 items), emotional blunting (17 items), and cognitive inertia (16 items), based on a Likert-type scale from 0 (no apathy) to 3 (severe apathy). This scale will be completed by a regular caregiver of the person with dementia, who in this case will be a professional at the site.
Agitation assessed through the Cohen-Mansfield Agitation Inventory (CMAI) | Baseline (T0)
  Cohen-Mansfield Agitation Inventory (CMAI). CMAI is a tool developed for the detection and assessment of agitation behavior in elderly people. The adaptation to Spanish of this tool is the Cohen-Mansfield Agitation Inventory of the elderly. In the same way as the APADEM-NH, this scale will be completed by a professional at the site who frequently works in the care of the user.
Change in agitation assessed through the Cohen-Mansfield Agitation Inventory (CMAI) | 12 weeks after the beginning of the intervention (T1)
  Cohen-Mansfield Agitation Inventory (CMAI). CMAI is a tool developed for the detection and assessment of agitation behavior in elderly people. The adaptation to Spanish of this tool is the Cohen-Mansfield Agitation Inventory of the elderly. In the same way as the APADEM-NH, this scale will be completed by a professional at the site who frequently works in the care of the user.
Change in agitation assessed through the Cohen-Mansfield Agitation Inventory (CMAI) | 12 weeks after end of the intervention (T2)
  Cohen-Mansfield Agitation Inventory (CMAI). CMAI is a tool developed for the detection and assessment of agitation behavior in elderly people. The adaptation to Spanish of this tool is the Cohen-Mansfield Agitation Inventory of the elderly. In the same way as the APADEM-NH, this scale will be completed by a professional at the site who frequently works in the care of the user.

OTHER OUTCOMES:
Psychotropic medication | Baseline (T0)
  Psychotropic medication (antidementia drugs, antidepressants, anxiolytics and antipsychotics) prescribed at baseline (T0)
Change in psychotropic medication | 12 weeks after the beginning of the intervention (T1)
  Change in psychotropic medication (antidementia drugs, antidepressants, anxiolytics and antipsychotics) prescribed between baseline (T0) and after the intervention (T1).
Rescue medication | 12 weeks after the beginning of the intervention (T1)
  Number of rescue medication doses used by each participant during the study period
Cost-Effectiveness | 12 weeks after the beginning of the intervention (T1)
  The cost-effectiveness measure will be the incremental cost-effectiveness ratio (ICER), obtained by dividing the difference between the cost of the PARO Therapy Robot intervention and the standard care by the difference in effectiveness (quality-adjusted life-years [QALY]) between the PARO Therapy Robot intervention and the standard care.
Acceptability of PARO robot | Post-intervention (T1) (after 12 weeks of robot therapy intervention)
  The technicians who have performed the intervention will complete a questionnaire to assess the acceptability of PARO with each user who has participated. The questionnaire comprises 7 items that assess the participants from the perspective of the therapists. The questionnaire to be used encompasses several aspects such as closeness to the robot, feeling of well-being during the interaction, practicality, and actions of rejection. Each item is scored on a Likert-type scale from 1-5, where 1 = totally disagree and 5 = totally agree.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Perez, Phd, Study Director — Centro de Referencia Estatal de atención a personas con enfermedad de Alzheimer y otras demencias - Imserso; Teresa Rodriguez, MSc, Principal Investigator — Centro de Referencia Estatal de atención a personas con enfermedad de Alzheimer y otras demencias - Imserso; Mireia Tofiño, MSc, Principal Investigator — Centro de Referencia Estatal de atención a personas con enfermedad de Alzheimer y otras demencias - Imserso
Locations (15):
- Spain (15):
  - ATENDO Calidade S.L, Vigo, Pontevedra
  - Centro Residencial CleceVitam Bastiagueiro, A Coruña
  - Residencia DomusVi Alcoi, Alicante
  - Residencia DomusVi Alicante Babel, Alicante
  - Residencia CleceVitam San Pedro Poveda, Burgos
  - Residencia DomusVi Vila-Real, Castelló
  - Residencia CleceVitam Ponent, Lleida
  - Residencia de Mayores Albertia Moratalaz, Madrid
  - Residencia ORPEA Madrid Buenavista, Madrid
  - Residencia ORPEA Pinto, Madrid
  - Centro Residencial CleceVitam Carmen Conde, Murcia
  - Residencia Bañosalud, Palencia
  - Residencia CleceVitam San Antonio, Salamanca
  - CleceVitam Gerohotel, Valladolid
  - Residencia León Trucíos, Vizcaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bemelmans R, Gelderblom GJ, Jonker P, de Witte L. Socially assistive robots in elderly care: a systematic review into effects and effectiveness. J Am Med Dir Assoc. 2012 Feb;13(2):114-120.e1. doi: 10.1016/j.jamda.2010.10.002. Epub 2010 Dec 15. PMID 21450215
- [Background] 2021 Alzheimer's disease facts and figures. Alzheimers Dement. 2021 Mar;17(3):327-406. doi: 10.1002/alz.12328. Epub 2021 Mar 23. PMID 33756057
- [Background] Asl AM, Toribio-Guzman JM, van der Roest H, Castro-Gonzalez A, Malfaz M, Salichs MA, Martin MF. The usability and feasibility validation of the social robot MINI in people with dementia and mild cognitive impairment; a study protocol. BMC Psychiatry. 2022 Dec 5;22(1):760. doi: 10.1186/s12888-022-04418-9. PMID 36471336
- [Background] Cohen-Mansfield J, Marx MS, Rosenthal AS. A description of agitation in a nursing home. J Gerontol. 1989 May;44(3):M77-84. doi: 10.1093/geronj/44.3.m77. PMID 2715584
- [Background] Frings L, Yew B, Flanagan E, Lam BY, Hull M, Huppertz HJ, Hodges JR, Hornberger M. Longitudinal grey and white matter changes in frontotemporal dementia and Alzheimer's disease. PLoS One. 2014 Mar 3;9(3):e90814. doi: 10.1371/journal.pone.0090814. eCollection 2014. PMID 24595028
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Kang HS, Makimoto K, Konno R, Koh IS. Review of outcome measures in PARO robot intervention studies for dementia care. Geriatr Nurs. 2020 May-Jun;41(3):207-214. doi: 10.1016/j.gerinurse.2019.09.003. Epub 2019 Oct 24. PMID 31668459
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Assessing quality of life in older adults with cognitive impairment. Psychosom Med. 2002 May-Jun;64(3):510-9. doi: 10.1097/00006842-200205000-00016. PMID 12021425
- [Background] Moniz-Cook E, Vernooij-Dassen M, Woods R, Verhey F, Chattat R, De Vugt M, Mountain G, O'Connell M, Harrison J, Vasse E, Droes RM, Orrell M; INTERDEM group. A European consensus on outcome measures for psychosocial intervention research in dementia care. Aging Ment Health. 2008 Jan;12(1):14-29. doi: 10.1080/13607860801919850. PMID 18297476
- [Background] Moyle W, Bramble M, Jones CJ, Murfield JE. "She Had a Smile on Her Face as Wide as the Great Australian Bite": A Qualitative Examination of Family Perceptions of a Therapeutic Robot and a Plush Toy. Gerontologist. 2019 Jan 9;59(1):177-185. doi: 10.1093/geront/gnx180. PMID 29165558
- [Background] O'Shea E, Devane D, Murphy K, Cooney A, Casey D, Jordan F, Hunter A, Murphy E. Effectiveness of a structured education reminiscence-based programme for staff on the quality of life of residents with dementia in long-stay units: a study protocol for a cluster randomised trial. Trials. 2011 Feb 14;12:41. doi: 10.1186/1745-6215-12-41. PMID 21320303
- [Background] Peters F, Villeneuve S, Belleville S. Predicting progression to dementia in elderly subjects with mild cognitive impairment using both cognitive and neuroimaging predictors. J Alzheimers Dis. 2014;38(2):307-18. doi: 10.3233/JAD-130842. PMID 23963293
- [Background] Pu L, Moyle W, Jones C. How people with dementia perceive a therapeutic robot called PARO in relation to their pain and mood: A qualitative study. J Clin Nurs. 2020 Feb;29(3-4):437-446. doi: 10.1111/jocn.15104. Epub 2019 Dec 2. PMID 31738463
- [Background] Martin Rico F, Rodriguez-Lera FJ, Gines Clavero J, Guerrero-Higueras AM, Matellan Olivera V. An Acceptance Test for Assistive Robots. Sensors (Basel). 2020 Jul 14;20(14):3912. doi: 10.3390/s20143912. PMID 32674372
- [Background] Saragih ID, Tonapa SI, Sun TL, Chia-Ju L, Lee BO. Effects of robotic care interventions for dementia care: A systematic review and meta-analysis randomised controlled trials. J Clin Nurs. 2021 Nov;30(21-22):3139-3152. doi: 10.1111/jocn.15856. Epub 2021 May 26. PMID 34041803
- [Background] Shibata T, Wada K. Robot therapy: a new approach for mental healthcare of the elderly - a mini-review. Gerontology. 2011;57(4):378-86. doi: 10.1159/000319015. Epub 2010 Jul 15. PMID 20639620
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Yu C, Sommerlad A, Sakure L, Livingston G. Socially assistive robots for people with dementia: Systematic review and meta-analysis of feasibility, acceptability and the effect on cognition, neuropsychiatric symptoms and quality of life. Ageing Res Rev. 2022 Jun;78:101633. doi: 10.1016/j.arr.2022.101633. Epub 2022 Apr 21. PMID 35462001
- [Background] Agüera-Ortiz L, Cruz-Orduña I, Ramos-García MI, Valentí-Soler, M, Gil-Ruiz N, Osorio-Suárez RM, Dobato JL, Olazarán-Rodríguez J, León-Salas B, Martínez-Martín P. Proceso de creación de la escala APADEM-NH para la medición de la apatía en pacientes con demencia institucionalizados. Psicogeriatría. 2011; 3: 29-36.
- [Background] Cervilla J, Rodríguez A, Hoyos G, Mínguez L, González E. Agitación y deterioro cognitivo usando la versión española del Inventario de agitación del anciano de Cohen-Mansfield. Psiquiatria.com-Revista internacional online. 2002; 6(5): 1-10.
- [Background] Glick HA, Doshi JA, Sonnad SS, Polsky D. Economic evaluation in clinical trials. 1st. ed. Oxford: Oxford University Press; 2007.
- [Background] Gomez-Gallego M, Gomez-Amor J, Gomez-Garcia J. [Validation of the Spanish version of the QoL-AD Scale in alzheimer disease patients, their carers, and health professionals]. Neurologia. 2012 Jan;27(1):4-10. doi: 10.1016/j.nrl.2011.03.006. Epub 2011 May 12. Spanish. PMID 21570161
- [Background] Inoue T, Nihei M, Narita T, Onoda M, Ishiwata R, Mamiya I, Shino M, Kojima H, Ohnaka S, Fujita Y, Kamata M. Field-based development of an information support robot for persons with dementia. Technology and Disability. 2012; 24(4): 263-271. doi: 10.3233/TAD-120357.
- [Background] Khosla R, Nguyen K, Chu MT. Human robot engagement and acceptability in residential aged care. International Journal of Human-Computer Interaction. 2017; 33(6): 510-522. doi: 10.1080/10447318.2016.1275435.
- [Background] Kolling T, Haberstroh J, Kaspar R, Pantel J, Oswald F, Knopf M. Evidence and deployment-based research into care for the elderly using emotional robots: psychological, methodological and cross-cultural facets. GeroPsych: The Journal of Gerontopsychology and Geriatric Psychiatry. 2013; 26(2): 83-88. doi: 10.1024/1662-9647/a000084.
- [Background] Logsdon RG, Gibbons LE, McCurry SM, Teri L. Quality of life in Alzheimer's disease: patient and caregiver reports. Journal of Mental Health and Aging. 1999; 5(1): 21-32.
- [Background] Martinez de la Iglesia J, Onis Vilches MC, Duenas Herrero R, Aguado Taberne C, Albert Colomer C, Arias Blanco MC. [Abbreviating the brief. Approach to ultra-short versions of the Yesavage questionnaire for the diagnosis of depression]. Aten Primaria. 2005 Jan;35(1):14-21. doi: 10.1157/13071040. Spanish. PMID 15691450
- [Background] Martínez-Velásquez DA, Chavarro-Carvajal DA, García-Cifuentes E, Venegas-Sanabria LC, Cano-Gutiérrez CA. Caracterización de pacientes con demencia avanzada hospitalizados por el servicio de geriatría en un hospital de alta complejidad. Acta Neurológica Colombiana. 2019; 35(1): 15-21. doi: 10.22379/24224022228.
- [Background] Moyle W, Jones C, Sung B, Bramble M, O'Dwyer S, Blumenstein M, Estivill-Castro V. What effect does an animal robot called CuDDler have on the engagement and emotional response of older people with dementia? A pilot feasibility study. International Journal of Social Robotics. 2016; 8(1): 145-156. doi: 10.1007/s12369-015-0326-7.
- [Background] Olazaran J, Reisberg B, Clare L, Cruz I, Pena-Casanova J, Del Ser T, Woods B, Beck C, Auer S, Lai C, Spector A, Fazio S, Bond J, Kivipelto M, Brodaty H, Rojo JM, Collins H, Teri L, Mittelman M, Orrell M, Feldman HH, Muniz R. Nonpharmacological therapies in Alzheimer's disease: a systematic review of efficacy. Dement Geriatr Cogn Disord. 2010;30(2):161-78. doi: 10.1159/000316119. Epub 2010 Sep 10. PMID 20838046
- [Background] Plan integral de Alzheimer y otras demencias (2019-2023). Madrid: Ministerio de Sanidad, Consumo y Bienestar Social; 2019.
- [Background] Shankar KK, Walker M, Frost D, Orrell MW. The development of a valid and reliable scale for rating anxiety in dementia (RAID). Aging & Mental Health. 1999; 3(1): 39-49. doi: 10.1080/13607869956424.
- [Background] Sheikh JI, Yesavage, JA. Geriatric Depression Scale (GDS): recent evidence and development of a shorter version. Clinical Gerontologist. 1986; 5: 165-73. doi: 10.1300/J018v05n01_09.
- [Background] Shibata T, Kawaguchi Y, Wada K. Investigation on people living with seal robot at home. International journal of social robotics. 2012; 4(1): 53-63. doi:10.1007/s12369-011-0111-1.